CLINICAL TRIAL: NCT06314815
Title: Ilioinguinal-iliohypogastric Nerve Block Prior to Shouldice Inguinal Hernia Repair
Acronym: NBSS
Status: Completed | Type: Observational
Sponsor: Shouldice Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Shouldice hospital
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Inguinal Hernia; Pain, Postoperative
Keywords: Inguinal hernia; Pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients that received the ilioinguinal-iliohypogastric nerve block [IINB] were chosen by the anesthetists prior to surgery based on patient suitability, consultation with patients, and availability of time and resources. The Ilioinguinal-iliohypogastric nerve block contained one of 0.5% Bupivacaine and 2% Lidocaine, 0.5% Marcaine and 2% Lidocaine, 0.25% Marcaine with Epinephrine, 0.25% or 0.1% Bupivacaine 2ith 2% Lidocaine (mixtures such as: 0.5% Bupivacaine (also called Marcaine) and 2% Lidocaine, with or without Epinephrine mix).
- 2: Matched patients in terms of biometric and peroperative data, who did not receive an Ilioinguinal-iliohypogastric nerve block.

SUMMARY:
The introduction of ilioinguinal-iliohypogastric nerve blocks into the preoperative care regimen at Shouldice Hospital for inguinal hernia repair marks a significant shift in pain management strategies. While Shouldice Hospital has traditionally not employed this technique, recent literature highlighting its potential benefits has prompted its trial within their patient population.

Research in this area, although limited, suggests promising outcomes. Studies such as those by Beaussier et al. (2005) and Nehra et al. (1995) have demonstrated decreased postoperative pain and opioid use, as well as increased mobility associated with the use of ilioinguinal-iliohypogastric nerve blocks. However, concerns such as orthostatic hypotension and rebound pain have also been noted, indicating the need for careful consideration and monitoring of potential adverse effects.

More recent studies, particularly those focusing on the Lichtenstein repair, have further supported the potential benefits of ilioinguinal-iliohypogastric nerve blocks. Kacmaz and Bolat (2020) found improved patient satisfaction, reduced opioid consumption, and shorter hospital stays associated with nerve block techniques. Additionally, the use of adjuncts such as dexamethasone has shown promise in reducing rebound pain and opioid requirements postoperatively.

The purpose of evaluating the use of ilioinguinal-iliohypogastric nerve blocks at Shouldice Hospital is multifaceted. Not only does it aim to enhance patient care and satisfaction by improving pain management strategies, but it also provides valuable insights for anesthetists and surgeons regarding the utility and efficacy of this technique within the context of inguinal hernia repair. Furthermore, the trial may facilitate the refinement of current practices, potentially leading to standardized protocols that optimize patient outcomes while minimizing adverse effects.

In summary, the introduction of ilioinguinal-iliohypogastric nerve blocks at Shouldice Hospital represents a proactive approach toward enhancing perioperative care for inguinal hernia patients. By leveraging emerging evidence and adapting to evolving clinical practices, the hospital stands to benefit from improved patient outcomes and potentially contribute to the advancement of pain management strategies in hernia surgery.

DETAILED DESCRIPTION:
Routine preoperative care at Shouldice Hospital has not classically included the use of an ilioinguinal-iliohypogastric nerve block. However, with the purchase of an ultrasound machine and growing reports in the literature to the benefit of nerve blocks for inguinal hernia surgery1-5, it is now being trialed in patients at Shouldice Hospital.

There is limited research on the outcomes of ilioinguinal-iliohypogastric nerve block for inguinal hernia patients undergoing a Shouldice Repair, and none from the Shouldice Hospital, founder of the repair. One of the few reports evaluated patients who underwent a modified Shouldice Technique and not the actual repair2. Beaussier et al (2005), reported on 40 patients, 20 received local anesthesia with an ilioinguinal-iliohypogastric nerve block and 20 just received local anesthesia, and measured time to first analgesic request, pain intensity, and adverse events2. Their findings showed that the ilioinguinal-iliohypogastric nerve block with local anesthesia group had less pain during movement on postoperative day 3 but had an increased risk for orthostatic hypotension2. An even earlier study by Nehra et al (1995), divided 200 male inguinal hernia patients, who underwent a Shouldice Technique or modified Bassini repair, into 4 different treatment groups for comparison1. The groups included bupivacaine ilioinguinal field block with oral aspirin, bupivacaine ilioinguinal field block with oral placebo, saline with oral aspirin, and saline with oral placebo1. They measured pain scores, mobility, complications, patient experience, as well as opioid use1. The authors found that the bupivacaine ilioinguinal field block with oral aspirin group had decreased pain and opioid use, as well as increased mobility compared to groups that had saline with oral aspirin and saline with oral placebo1.

More recent research, focusing exclusively on the Lichtenstein repair for inguinal hernias, found that treatment groups had improved outcomes4,5. Kacmaz and Bolat (2020), compared 35 patients who received spinal anesthesia with 35 who received an ilioinguinal-iliohypogastric nerve block with tumescent anesthesia4. They measured sensory block onset time, patient satisfaction, postoperative opioid consumption, duration of surgery and first mobilization, length of hospital stay due to complications related to anesthetic method, and intraoperative hemodynamic values4. The authors found that in the nerve block group there was an increased duration of sensory block, intraoperative pain scores, and patient satisfaction, as well as lower postoperative pain scores, need for analgesics, and urinary retention, there was also early mobilization and discharge4. A 2023 study comparing 30 patients who received an ilioinguinal-iliohypogastric nerve block with added dexamethasone to 30 who just received a nerve block, found that the combination group had decreased rebound pain scores and opioid use5.

The purpose of this study is to evaluate the use of ilioinguinal-iliohypogastric nerve block for hernia patients at Shouldice Hospital. The results are expected to be useful in implementing the ilioinguinal-iliohypogastric nerve block within the patient population at Shouldice Hospital. Concurrently, aiding in understanding and potentially improving the current practices regarding pain management. This could enhance patient care and satisfaction, as well as provide valuable information about the utility of an ilioinguinal-iliohypogastric nerve block to the anesthetists and surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all gender
* Shouldice repair due to a groin hernia operation at Shouldice Hospital.

Exclusion Criteria:

* Missing information in patient charts or patients are unable to be matched 1:1

Ages: 16 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population will focus on all patients that had a hernia operation at Shouldice Hospital. The exclusion criteria are if there is missing information in patient charts or patients are unable to be matched 1:1. As this is the first study of its kind at Shouldice Hospital the required sample size is unknown, and we intend to include a small pilot analysis.
  The patients that receive the ilioinguinal-iliohypogastric nerve block are having it administered in the operating room when on the table. The onset of the block is within minutes and lasts up to 12 hours after administration. The ilioinguinal-iliohypogastric nerve block is an option for almost everyone and may provide additional support for patients with lower pain thresholds and/or substance use issues. There is no difference in postoperative course for those patients who do and do not receive the nerve block, and there are no additional risks.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Compare pain and pain medication use between patients receiving an ilioinguinal-iliohypogastric nerve block prior to hernia surgery with those who do not. | 3 days after surgery
  Aldrete scoring/system

SECONDARY OUTCOMES:
Evaluate the impact of the ilioinguinal-iliohypogastric nerve block on patients with pain conditions, mental health conditions, and substance use histories. | 3 days after surgery
  Aldrete scoring/system
Determine sample size for future prospective trial. | 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite Mainprize, Principal Investigator — Shouldice Hospital
Locations (1):
- Shouldice hospital, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1- Nehra D, Gemmell L, Pye JK. Pain relief after inguinal hernia repair: a randomized double-blind study. Br J Surg. 1995;82(9):1245-7. https://doi.org/10.1002/bjs.1800820929 2- Beaussier M, Weickmans H, Abdelhalim Z, Lienhart A. Inguinal herniorrhaphy under monitored anesthesia care with ilioinguinal-iliohypogastric block: the impact of adding clonidine to ropivacaine. Anesth Analg. 2005;101(6):1659-62. https://doi.org/10.1213/01.ANE.0000184046.64631.50 3- Stav A, Reytman L, Stav MY, Troitsa A, Kirshon M, Alfici R, Dudkiewicz M, and Sternberg A. Transversus abdominis plane versus ilioinguinal and iliohypogastric nerve blocks for analgesia following open inguinal herniorrhaphy. Rambam Maimonides Medical Journal. 2016;7(3). 4- Kacmaz M and Bolat H. Comparison of spinal anaesthsia versus ilioinguinal-iliohypogastric nerve block applied with tumescent anaesthsia for single-sided inguinal hernia. Hernia. 2020;24;1049-1056. 5- Korkusuz M, Basaran B, Et T, Bilge A, Yarimoglu R, and Kurucay Y. The effects of dexamethasone added to ilioinguinal/iliohypogastric nerve (IIN/IHN) block on rebound pain in inguinal hernia surgery: a randomized controlled trial. Hernia. 2023. https://doi.org/10.1007/s10029-023-02841-9.